CLINICAL TRIAL: NCT06531486
Title: A Multicenter, Open Label, Single-arm Phase I/II Dose-escalation and Dose-expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, and Initial Efficacy of XS-02 Capsules in Patients With Advanced Solid Tumors
Brief Title: A Study of XS-02 Capsules in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NovaOnco Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XS-02-I101
Record Dates: First submitted 2024-05-28; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Solid Tumor; Ovarian Cancer; Breast Cancer; Endometrial Cancer
Keywords: XS-02; Cell cycle checkpoint kinase 1（CHK1); Solid tumor; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase I dose escalation/Phase II dose expansion (Experimental): Experimental: XS-02 Dosage form:capsule Specification: 5mg，25mg Dose: Phase I dose escalation, orally, once daily, the administration schedule (including dose,administration frequency/interval, administration cycle, etc.) can be adjusted according to the experimental data. Phase II Dose Expansion/Optimal Dose selection, will be determined based on the Phase I dose escalation results.
  Method of administration: Oral
  Interventions: Other: XS-02 capsules

INTERVENTIONS:
Other: XS-02 capsules — Upon completion of all screening visits, eligible patients will be treated with XS-02 capsules at the appropriate dose.

SUMMARY:
A study to evaluate the safety, tolerability, Pharmacokinetics(pk), and efficacy of XS-02 capsules in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a multicenter, open label, single-arm Phase I/II dose-escalation and dose-expansion study to evaluate the safety, tolerability, pharmacokinetic profile, and initial efficacy of XS-02 capsules in patients with advanced solid tumors.

ELIGIBILITY:
inclusion criteria:

* Volunteer to participate in clinical trials and sign an informed consent form (ICF).
* Age ≥18 years old, ≤75 years old, regardless of gender.
* Patients with locally advanced or metastatic solid tumors diagnosed histologically or cytologically have no standard treatment options or have failed standard treatment or are unable to tolerate standard treatment. Phase II dose expansion/Optimal dose selection phase enrolls advanced ovarian cancer and other advanced entities a tumor patient.
* The phase I dose escalation phase has at least one evaluable lesion and the phase II dose expansion/optimal dose selection phase has at least one measurable lesion (based on RECIST V1.1). For patients who have previously received radiation therapy, a radiation-treated lesion may be considered a target lesion if the lesion can be measured according to RECIST V1.1 and there is objective evidence of significant progression after radiation therapy.
* The Eastern Cooperative Oncology Group (ECOG) scored 0-1.
* The expected survival time is ≥3 months.
* Routine blood tests before first dosing must be within the following range (no blood transfusion or use of drugs that assist in raising white blood cells, platelets, hemoglobin, such as cytokines or erythropoietin, etc., for at least 7 days prior to first dosing)

  1. Hemoglobin (HB) ≥90 g/L.
  2. Platelet (PLT) count ≥100×109/L or ≥5.6 mmol/L.
  3. Absolute count of neutrophils (ANC) ≥1.5×109/L.
* Has proper organ function
* Female subjects of reproductive age in the screening period had negative serological pregnancy test results within 7 days prior to the first dosing. The subjects also agreed to use a reliable method of contraception for 3 months from signing the informed consent to the last dosing. Including but not limited to: forbidden Sex, male vasectomy, female sterilization, effective IUD, condoms, effective contraceptive drugs.
* Patients were able to comply with the visits required by the study procedure and protocol.

Admission criteria specific to Stage II dose expansion/Optimal dose Selection stage ovarian cancer:

* Histologically confirmed and documented advanced recurrent epithelial ovarian cancer (high-grade serous ovarian cancer), fallopian tube cancer, and primary peritoneal cancer.
* For platinum-resistant diseases, there must be evidence of disease progression within 6 months of the most recent platinum-containing treatment, calculated from the date of the last platinum treatment dose. Platinum-refractory patients were not admitted (platinum-refractory was defined as during or after chemotherapy containing platinum-containing chemotherapy)Progress within 4 weeks.
* Have previously received at least 1 standard line of treatment.

exclusion criteria:

* Chemotherapy, small molecule targeted therapy, endocrine therapy and traditional Chinese medicine with anti-tumor indications were received within 2 weeks prior to the first dose. Received tumor immunotherapy, antibodies, polypeptide antitumor, or other investigational drugs within 4 weeks prior to initial administration.
* Patients who had undergone therapeutic surgery other than diagnosis, biopsy, drainage, or radical radiotherapy within 4 weeks prior to initial dosing, or who expected to undergo major surgery during the study period. Had received palliative radiotherapy within 2 weeks prior to the first dose, or had used radiopharma (strontium, samarium, etc.) within 56 days prior to the first dose.
* The toxicity of previous antitumor therapy has not recovered (> NCI-CTCAE 5.0 grade 1),alopecia, pigmentation, or other toxicity that the investigators assessed had become chronic and did not affect the safety of the investigational medication returned to NCI-CTCAE 5.0 level 2 or below.
* Imaging (Computed Tomography(CT) or magnetic resonance imaging(MRI)) shows that the tumor has invaded large blood vessels (such as aorta, pulmonary artery, pulmonary vein, vena cava, etc.) or is at risk of bleeding (such as esophageal and gastric varices).
* inflammatory breast cancer
* There is clinically uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage or medical intervention (within 2 weeks prior to administration).
* Patients with central nervous system metastasis who meet any of the following conditions:

  1. need to undergo local treatment (surgery, radiation or other);
  2. Patients who require steroid hormones, anticonvulsants, or other dehydration treatment;
  3. Only enrollment is allowed Stable symptoms, imaging assessment (imaging evaluation of brain metastases within 4 weeks prior to enrollmentlesions that have not progressed) and do not require treatment
* Patients with difficulty swallowing, or a history of severe gastrointestinal disease (e.g. active inflammatory bowel disease, gastrointestinal perforation) and related symptoms that cannot be reasonably controlled; Or have a gastrointestinal disorder (e.g., Crohn's disease, ulcerative colitis, intestinal obstruction, short bowel syndrome) or other malabsorption conditions that affect drug absorption.
* Have active or unstable cardiovascular disease
* Bacterial, fungal, or viral infections requiring intravenous antibiotics/antivirals or hospitalization were investigated within 2 weeks prior to initial drug administration.
* People who have a history of prior severe allergies, or are allergic to any active or inactive ingredient of the investigatory drug.
* Known acute or active hepatitis B (hepatitis B virus（HBV） surface antigen positive with HBV deoxyribonucleic acid（DNA）≥500 IU/mL), hepatitis C virus infection (HCV Ribonucleic Acid（RNA） exceeding the normal range), syphilis infection, and human immunodeficiency virus (HIV) infection.
* Other primary malignancies have been diagnosed within the previous five years (the following conditions can be included: cured and completely resected basal and squamous cell skin cancers, completely resected cancers of any type in situ).
* Use within 2 weeks prior to first administration, or expect to use a Cytochrome P450 enzyme(CYP3A) booster or strong inducer during study drug administration.
* Use within 2 weeks prior to first administration, or expect to use any drug known to prolong the corrected QT(QTc) interval during study drug administration.
* The ATR/CHK1 pathway has been treated in the past.
* Had a bone marrow transplant or had extensive radiation therapy on more than 25% of the bone marrow in the 8 weeks prior to initial dosing.
* A history of blood clotting disorders; Anticoagulant or antiplatelet therapy (oral aspirin dose ≤100 mg/d and subcutaneous injection of low molecular weight heparin for prevention of deep vein thrombosis) is required.
* Pregnant and lactating women.
* According to the judgment of the investigator, any other serious or uncontrolled acute or chronic diseases or abnormal laboratory tests or other reasons are not suitable for participation in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-07-29 (Estimated); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicity (DLT) (DLT observation period).(phase I) | from first dose up to 31 days
  DLT is defined as a dose-limiting toxic event that occurs during DLT observation.
Maximum tolerated dose (MTD) and/or Recommended Phase II Dose(RP2D).(phase I) | Time Frame: from first dose to phase I completion, an average of 1.5 years
  MTD is defined as the maximum tolerated dose。RP2D is defined as the recommended dose for Phase II clinical studies
Objective Response Rate（ORR）(phase II) | Through study completion, an average of 3 years
  ORR is defined as the proportion of patients with confirmed Complete Response (CR) or Partial Response (PR) as evaluated according to RECIST version 1.1.

SECONDARY OUTCOMES:
the incidence and severity of adverse events, serious adverse events, deaths, and safety screening abnormalities(phase I/II) | From enrollment up to 30 days after last dose
  According to National Cancer Institute Common Terminology Criteria for Adverse Events(NCI-CTCAE) version 5.0 evaluates the incidence and severity of adverse events, serious adverse events, deaths, and safety screening abnormalities (such as laboratory tests, vital signs, physical examinations, electrocardiograms, ECOG, etc.). Proportion of patients undergoing dose adjustment or discontinuation due to drug toxicity.
Pharmacokinetics(PK) parameters(phase I/II) | up to 12 weeks
  Area under the concentration-time curve from time 0 (pre-dose) to the last measurable time of concentration(AUC0-t)
PK parameters(phase I/II) | up to 12 weeks
  Area under the concentration-time curve from time 0 (pre-dose) to infinity(AUC0-∞)
PK parameters(phase I/II) | up to 12 weeks
  Area under the plasma drug concentration-time curve over a dosing interval at steady state(AUCtau)
PK parameters(phase I/II) | up to 12 weeks
  Maximum plasma concentration(Cmax)
PK parameters(phase I/II) | up to 12 weeks
  Time to maximum plasma concentration(Tmax)
PK parameters(phase I/II) | up to 12 weeks
  half-life(t1/2)
Disease Control Rate(DCR)(phase I/II) | Through study completion, an average of 3 years
  DCR is defined as the proportion of patients with confirmed Complete Response(CR), Partial Response(PR), and Stable Disease(SD) based on the Response Evaluation Criteria in Solid Tumors Version 1.1(RECISIT V1.1) evaluation.
（Clinical Benefit Rate(CBR)(phase I/II) | Through study completion, an average of 3 years
  CBR was defined as the proportion of patients with CR, PR, and SD lasting at least 24 weeks, as evaluated according to RECIST version 1.1.
Duration of Response（DOR）(phase I/II) | Through study completion, an average of 3 years
  DOR is defined as the time from the date of first documented response (which is subsequently confirmed) until progression per RECIST V1.1 criteria or death due to any cause
Time to Response（TTR）(phase I/II) | Through study completion, an average of 3 years
  TTR is defined as the time from the first dose to the first confirmed PR or CR evaluated according to RECIST version 1.1.
Progression Free Survival（PFS）(phase I/II) | Through study completion, an average of 3 years
  PFS is defined as the time until disease progression or death of the first dose, whichever occurs first.
Overall Survival（OS）(phase I/II) | Through study completion, an average of 3 years
  OS is defined as the time from the first use of the study drug until death from any cause.
Objective Response Rate（ORR）(phase I) | from first dose to phase I completion, an average of 1.5 years
  ORR is defined as the proportion of patients with confirmed Complete Response (CR) or Partial Response (PR) as evaluated according to RECIST version 1.1.

IPD SHARING:
Plan to Share IPD: No